CLINICAL TRIAL: NCT04405193
Title: The Efficacy of N-acetylcysteine Versus Placebo for the Treatment of Metamphetamine Withdrawal Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Melva Louisa (Other)
Responsible Party: Sponsor-Investigator, Melva Louisa, Dr Melva Louisa, SSi, MBiomed; Research Coordinator for the Department of Pharmacology and Therapeutics, Primary Investigator, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UI-BNN
Record Dates: First submitted 2020-04-21; First posted 2020-05-28 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Methamphetamine Dependence in Remission
Keywords: methamphetamine; N-acetylcysteine; substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Randomised, parallel, 4 week-treatment of N-acetylcysteine versus matching placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 2 capsules, each containing 600 mg N-acetylcysteine administered once daily every morning.
  Interventions: Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): 2 capsules of matching placebo administered once daily every morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetyl cysteine — Eligible patients will be randomised to receive N-acetylcysteine or placebo
  Other Names: Placebo
  Arms: Treatment
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
Up to date, no approved medications are available for the treatment of methamphetamine addiction. Recently, N-acetylcysteine is recently being studied for methamphetamine withdrawal.

N-acetylcysteine, is a drug that has been long used as a mucolytic. Recent studies investigate the use of N-acetylcysteine in cocaine and withdrawal symptoms by its effect on restoring glutamate homeostasis in nucleus accumbens. Up to date, there has been 2 pilot study investigating the efficacy of N-acetylcysteine for methamphetamine dependence.

The present study is aimed to confirm the efficacy and safety of N-acetylcysteine in the treatment of methamphetamine withdrawal symptoms.

DETAILED DESCRIPTION:
Methamphetamine is a stimulant commonly abused worldwide. Methamphetamine can produce a rapid pleasurable rush caused by release of dopamine, nor-ephinephrine and serotonin. It produces euphoria, a heightened level of alertness and increased level of alertness and increased energy. Long-term regular meth use can lead to severe tooth decay, infection, weight loss, malnutrition, kidney damage, liver damage, respiratory issues, paranoia, violent behaviour, psychosis, severe anxiety and depression.

Studies suggested that withdrawal symptoms in methamphetamine dependent patients were due to the state of hypodopaminergic activities.

Up to date, no approved medications are available for the treatment of methamphetamine addiction. Recently, N-acetylcysteine is recently being studied for methamphetamine withdrawal.

N-acetylcysteine, is a drug that has been long used as a mucolytic. Up to date, there has been 2 pilot study investigating the efficacy of N-acetylcysteine for methamphetamine dependence. The present study is aimed to confirm the efficacy and safety of N-acetylcysteine in the treatment of methamphetamine withdrawal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 - 60 years old
* Diagnosed with methamphetamine addiction based on DSM-V criteria, enrolling for methamphetamine withdrawal treatment
* Agree to participate in the trial by signing informed consent

Exclusion Criteria:

* Known hypersensitivity to N-acetylcysteine
* Patients with serious conditions that will not allow protocol compliance or safe participation in the clinical trials.
* Pregnant or breastfeeding women
* History of suicidal thoughts / behaviour
* History of N-acetylcysteine treatment
* History of asthma and convulsions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Methamphetamine withdrawal symptoms in patients treated with N-acetylcysteine vs placebo | Change from baseline at 1 week.
  Withdrawal symptoms will be measured using Addiction Severity Index (ASI). ASI score ranged from 0 to 9, with score of 0 indicates no withdrawal symptoms and 9 indicates extreme symptoms of withdrawal symptoms
Methamphetamine withdrawal symptoms in patients treated with N-acetylcysteine vs placebo | Change from baseline at 2 weeks
  Withdrawal symptoms will be measured using Addiction Severity Index (ASI). ASI score ranged from 0 to 9, with score of 0 indicates no withdrawal symptoms and 9 indicates extreme symptoms of withdrawal symptoms
Methamphetamine withdrawal symptoms in patients treated with N-acetylcysteine vs placebo | Change from baseline at 4 weeks
  Withdrawal symptoms will be measured using Addiction Severity Index (ASI). ASI score ranged from 0 to 9, with score of 0 indicates no withdrawal symptoms and 9 indicates extreme symptoms of withdrawal symptoms

SECONDARY OUTCOMES:
Antioxidative effects of N-acetylcysteine vs placebo | Change from baseline at 4 weeks
  antioxidative effects will be measured by quantifying malondialdehyde plasma concentrations (micromol/L).
Safety of N-acetylcysteine vs placebo | Subjects with adverse events at week 1
  The number of subjects with adverse events at week 1
Safety of N-acetylcysteine vs placebo | Subjects with adverse events at week 2
  The number of subjects with adverse events at week 2
Safety of N-acetylcysteine vs placebo | Subjects with adverse events at week 4
  The number of subjects with adverse events at week 4

CONTACTS AND LOCATIONS:
Overall Officials: Erniawati Lestari, MD, Study Chair — Indonesia University
Locations (1):
- Rehabilitation Center, National Narcotics Agency, Bogor, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The results will be published in peer-reviewed journal

REFERENCES:
- [Background] Ling W, Mooney L, Haglund M. Treating methamphetamine abuse disorders. Curr Psychiatry. 2014; 13(9): 37 - 44.
- [Background] Winslow BT, Voorhees KI, Pehl KA. Methamphetamine abuse. Am Fam Physician. 2007 Oct 15;76(8):1169-74. PMID 17990840
- [Background] Prakash MD, Tangalakis K, Antonipillai J, Stojanovska L, Nurgali K, Apostolopoulos V. Methamphetamine: Effects on the brain, gut and immune system. Pharmacol Res. 2017 Jun;120:60-67. doi: 10.1016/j.phrs.2017.03.009. Epub 2017 Mar 14. PMID 28302577
- [Background] Ballester J, Valentine G, Sofuoglu M. Pharmacological treatments for methamphetamine addiction: current status and future directions. Expert Rev Clin Pharmacol. 2017 Mar;10(3):305-314. doi: 10.1080/17512433.2017.1268916. Epub 2016 Dec 20. PMID 27927042
- [Background] McKetin R, Dean OM, Baker AL, Carter G, Turner A, Kelly PJ, Berk M. A potential role for N-acetylcysteine in the management of methamphetamine dependence. Drug Alcohol Rev. 2017 Mar;36(2):153-159. doi: 10.1111/dar.12414. Epub 2016 May 30. PMID 27241765
- [Background] Nocito Echevarria MA, Andrade Reis T, Ruffo Capatti G, Siciliano Soares V, da Silveira DX, Fidalgo TM. N-acetylcysteine for treating cocaine addiction - A systematic review. Psychiatry Res. 2017 May;251:197-203. doi: 10.1016/j.psychres.2017.02.024. Epub 2017 Feb 11. PMID 28213190
- [Background] Grant JE, Odlaug BL, Kim SW. A double-blind, placebo-controlled study of N-acetyl cysteine plus naltrexone for methamphetamine dependence. Eur Neuropsychopharmacol. 2010 Nov;20(11):823-8. doi: 10.1016/j.euroneuro.2010.06.018. Epub 2010 Jul 22. PMID 20655182
- [Background] Mousavi SG, Sharbafchi MR, Salehi M, Peykanpour M, Karimian Sichani N, Maracy M. The efficacy of N-acetylcysteine in the treatment of methamphetamine dependence: a double-blind controlled, crossover study. Arch Iran Med. 2015 Jan;18(1):28-33. PMID 25556383